CLINICAL TRIAL: NCT06195982
Title: Acute Effects of Ketones in Heart Failure With Reduced Ejection Fraction
Brief Title: Ketones in Heart Failure With Reduced Ejection Fraction
Acronym: HFrEF
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00111539; 1K23HL161348-01 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-01-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; ketones; ketosis; metabolism; exercise
MeSH Terms: conditions — Heart Failure; Ketosis; Motor Activity | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Overview: The overall study design will be a randomized, double-blind crossover comparison of ketone ester (KE) therapy vs. KE-free vehicle in 25 patients with established HF with reduced ejection fraction (HFrEF). The main outcomes will be measures of exercise performance (peak and submaximal exercise).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ketone ester (Experimental): (R)-3-hydroxybutyl (R)-3-hydroxybutyrate, a ketone ester
  Interventions: Dietary Supplement: ketone ester
- placebo (Placebo Comparator): KE-free solution
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ketone ester — 500 mg/kg of ketone ester administered approximately 1 hour prior to the maximal exercise testing and 250 mg/kg administered approximately 30 minutes prior to submaximal exercise testing
  Other Names: ketone drink; KE drink; KE therapy; DeltaG therapy; ketone therapy
  Arms: ketone ester
Dietary Supplement: placebo — ketone-free placebo administered approximately 1 hour prior to the maximal exercise testing and ketone-free placebo administered approximately 30 minutes prior to submaximal exercise testing
  Arms: placebo

SUMMARY:
The purpose of this study is to understand the effects of a ketone drink on exercise capacity and other cardiovascular parameters in patients with heart failure. In heart failure, patients are limited in their ability to do all the things they want to do, and exercise as much as they would like, due to becoming tired and short of breath early. There may be several reasons why these symptoms occur. This study is assessing whether the ketone drink can improve these symptoms. This drink has been given status by Food and Drug Administration as "generally regarded as safe".

The use of DeltaG in this study is experimental. DeltaG has not been approved by the Food and Drug Administration (FDA) for the use being evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Stable cardiovascular medical therapy for 2 weeks
2. Participants will be required to have heart failure with reduced ejection fraction (left ventricular EF </= 45%) and New York Heart Association (NYHA) class II or III symptoms. In cases of ambiguity of functional status, reduced peak VO2 (<85% predicted VO2) at the baseline visit can be used to confirm reduced exercise tolerance.

Exclusion Criteria:

1. Intentional ketogenic diet in the last week
2. Cirrhosis or significant alcohol consumption
3. Contraindications to stress testing, conditions that limit exercise, and other clinically-significant causes of exertional limitation (claudication with peripheral artery disease, atrial fibrillation and heart rate >110 at rest, systolic blood pressure>180 mmHg or diastolic blood pressure>110 mmHg, infiltrative/hypertrophic cardiomyopathy, clinically significant pericardial disease, joint or neuromuscular disease that precludes exercise, acute coronary syndrome within the last 2 months, estimated glomerular filtration rate<20 mL/min/1.73 m2, and hemoglobin < 9 mg/dL).
4. Clinically significant lung disease: supplemental oxygen (aside from obstructive sleep apnea), chronic obstructive pulmonary disease requiring home oxygen or exacerbation within the last 2 months requiring steroids or antibiotics, severe obstructive lung disease (Gold stage 3).
5. >/= Moderate aortic stenosis, >mild mitral stenosis, > moderate aortic or mitral regurgitation
6. Type 1 diabetes mellitus
7. Implant of cardiac resynchronization therapy, cardiac contractility modulation, or barostim device within the previous 3 months.
8. Systolic blood pressure <90 mmHg
9. Pregnant women
10. Angina due to epicardial coronary disease or known presence of clinically-significant, unrevascularized epicardial coronary disease, in the investigator's opinion.
11. History of heart transplant, left ventricular assist device, or use of inotropic medication.
12. Participation in another clinical study with an investigational product in the previous 4 weeks prior to enrollment.
13. Conditions that may render the patient unable to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | 60 minutes after the intervention
  Peak VO2 assessed by cardiopulmonary exercise testing
Submaximal exercise capacity | 30 minutes after the intervention
  Exercise time at 75% of peak workload assessed by cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Left ventricular systolic function | Assessed 30 minutes after the intervention
  Left ventricular ejection fraction measured during resting echocardiography.
Substrate utilization | 60 minutes after the intervention
  Substrate utilization (reflected by the respiratory exchange ratio) assessed by cardiopulmonary exercise testing.
Left ventricular filling pressures | Assessed 60 minutes after the intervention
  E/e' ratio measured during stress echocardiography
Vasodilation at rest | 60 minutes after the intervention
  Total peripheral resistance measured at rest (calculated using cardiac output from echocardiography and brachial blood pressure)

OTHER OUTCOMES:
Right ventricular function | Assessed 30 minutes after the intervention
  Right ventricular function (tricuspid annular planar systolic excursion) assessed by echocardiography at rest
Cardiac output | Assessed 60 minutes after the intervention
  Cardiac output measured during stress echocardiography
Vasodilation during exercise | 60 minutes after the intervention
  Total peripheral resistance measured during cardiopulmonary exercise testing
Pulse wave velocity | Assessed 50 minutes after the intervention
  Pulse wave velocity measured by arterial tonometry
VO2 efficiency | Assessed 30 minutes after the intervention
  VO2 efficiency (total work performed over oxygen consumed) during submaximal cardiopulmonary exercise testing
Arterial stiffness | Assessed 50 minutes after the intervention
  Central augmentation index measured during arterial tonometry
Anaerobic threshold | Assessed 60 minutes after the intervention
  Anaerobic threshold measured during cardiopulmonary exercise testing
Pulmonary artery pressure | Assessed 60 minutes after the intervention
  Pulmonary artery systolic pressure assessed through echocardiography during cardiopulmonary exercise testing
Ventilatory efficiency | Assessed 60 minutes after the intervention
  VE/VCO2 measured during cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Selvaraj, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No